CLINICAL TRIAL: NCT04378166
Title: The Usefulness of Smart-glasses During Ultrasound-guided Central Venous Catheterization in Pediatric Patients: a Randomized Controlled Trial
Brief Title: AR for Pediatric Central Venous Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2003-018-1106
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: Compares central venous catheterization using smart-glasses and conventional method
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart glasses (Experimental): Application of smart glasses for ultrasound-guided central venous catheterization
  Interventions: Device: Smart glass
- Control (No Intervention): Conventional ultrasound-guided central venous catheterization

INTERVENTIONS:
Device: Smart glass — Practitioner wears smart glasses connected to ultrasound machine during central venous catheterization
  Arms: Smart glasses

SUMMARY:
This study is intended to investigate usefulness of smart-glasses for ultrasound-guided central venous catheterization in pediatric patients, by comparing success rate and elapsed time. The hypothesis is that smart-glasses would increase success rate in first trial.

DETAILED DESCRIPTION:
After obtaining informed consent from patients' legal guardian, children aged 6 or less undergoing surgery with need for central venous catheterization will be enrolled to the study.

Patients will be divided into either study group or control group. After anesthetic induction, central venous catheterization will be performed under ultrasound guidance. For patients in study group, the practitioner will be equipped with smart-glasses, while conventional ultrasound-guided catheterization will be performed for patients in control group.

Success rate of first trial, overall success rate, elapsed time during catheterization, complication regarding catheterization will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned to undergo surgery under general anesthesia
* Patients in need for central venous catheterization during anesthesia

Exclusion Criteria:

* Patients who have any of infection, hematoma, skin lesion, recent attempt of puncture at right internal jugular vein
* Patients with unstable vital sign prior to anesthetic induction
* Patients who are not eligible for catheterization at right internal jugular vein
* Refusal of legal guardian of patient

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
1st success rate | From start of central venous catheterization to successful placement of the guidewire at superior vena cava. Not to exceed 20 minutes.
  Success rate of central venous catheterization in first trial

SECONDARY OUTCOMES:
Overall success rate | From start of central venous catheterization to successful placement of the guidewire at superior vena cava. Not to exceed 3 attempts and 20 minutes.
  Overall success rate of central venous catheterization
Elapsed time for catheterization | From start of central venous catheterization to finish of catheterization. Not to exceed 3 attempts and 20 minutes.
  Overall elapsed time of central venous catheterization
Complication | From end of catheterization to 24 hours after catheterization
  Incidence and characteristics of complication related to central venous catheterization
Satisfaction score | From start of catheterization to end of catheterization. Not to exceed 20 minutes.
  5-points satisfaction score of practitioner (5 - Best / 4 - Good / 3 - Acceptable / 2 - Poor / 1 - Worst)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alderson PJ, Burrows FA, Stemp LI, Holtby HM. Use of ultrasound to evaluate internal jugular vein anatomy and to facilitate central venous cannulation in paediatric patients. Br J Anaesth. 1993 Feb;70(2):145-8. doi: 10.1093/bja/70.2.145. PMID 8435256
- [Background] Lau CS, Chamberlain RS. Ultrasound-guided central venous catheter placement increases success rates in pediatric patients: a meta-analysis. Pediatr Res. 2016 Aug;80(2):178-84. doi: 10.1038/pr.2016.74. Epub 2016 Apr 8. PMID 27057741
- [Background] Verghese ST, McGill WA, Patel RI, Sell JE, Midgley FM, Ruttimann UE. Comparison of three techniques for internal jugular vein cannulation in infants. Paediatr Anaesth. 2000;10(5):505-11. doi: 10.1046/j.1460-9592.2000.00554.x. PMID 11012954
- [Background] de Souza TH, Brandao MB, Nadal JAH, Nogueira RJN. Ultrasound Guidance for Pediatric Central Venous Catheterization: A Meta-analysis. Pediatrics. 2018 Nov;142(5):e20181719. doi: 10.1542/peds.2018-1719. PMID 30361397
- [Background] Hiranaka T, Nakanishi Y, Fujishiro T, Hida Y, Tsubosaka M, Shibata Y, Okimura K, Uemoto H. The Use of Smart Glasses for Surgical Video Streaming. Surg Innov. 2017 Apr;24(2):151-154. doi: 10.1177/1553350616685431. Epub 2017 Jan 9. PMID 28068887
- [Background] Huang CY, Thomas JB, Alismail A, Cohen A, Almutairi W, Daher NS, Terry MH, Tan LD. The use of augmented reality glasses in central line simulation: "see one, simulate many, do one competently, and teach everyone". Adv Med Educ Pract. 2018 May 10;9:357-363. doi: 10.2147/AMEP.S160704. eCollection 2018. PMID 29785148
- [Background] Rochlen LR, Levine R, Tait AR. First-Person Point-of-View-Augmented Reality for Central Line Insertion Training: A Usability and Feasibility Study. Simul Healthc. 2017 Feb;12(1):57-62. doi: 10.1097/SIH.0000000000000185. PMID 27930431
- [Background] Song IK, Kim EH, Lee JH, Jang YE, Kim HS, Kim JT. Seldinger vs modified Seldinger techniques for ultrasound-guided central venous catheterisation in neonates: a randomised controlled trial. Br J Anaesth. 2018 Dec;121(6):1332-1337. doi: 10.1016/j.bja.2018.08.008. Epub 2018 Sep 7. PMID 30442261
- [Background] Bruzoni M, Slater BJ, Wall J, St Peter SD, Dutta S. A prospective randomized trial of ultrasound- vs landmark-guided central venous access in the pediatric population. J Am Coll Surg. 2013 May;216(5):939-43. doi: 10.1016/j.jamcollsurg.2013.01.054. Epub 2013 Mar 7. PMID 23478546
- [Background] Song IK, Lee JH, Kang JE, Oh HW, Kim HS, Park HP, Kim JT. Comparison of central venous catheterization techniques in pediatric patients: needle vs angiocath. Paediatr Anaesth. 2015 Nov;25(11):1120-6. doi: 10.1111/pan.12726. Epub 2015 Aug 6. PMID 26248059